CLINICAL TRIAL: NCT00051077
Title: A Phase II Study of Adefovir Dipivoxil, Pegylated Interferon Alfa-2A, and Ribavirin Treatment in HBV and HCV Infected Subjects With HIV Disease
Brief Title: Treatment of Hepatitis in Patients Who Are Triple-Infected With HIV, Hepatitis B Virus (HBV), and Hepatitis C Virus (HCV)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: A5149; 10953 (Registry Identifier: DAIDS ES Registry Number); ACTG A5149
Record Dates: First submitted 2003-01-03; First posted 2003-01-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis B; Hepatitis C
Keywords: HIV Infections; Hepatitis B; Hepatitis C; Interferon Alfa-2a; Adefovir dipivoxil; Ribavirin; Antiviral Agents; Drug Resistance, Viral; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis C | interventions — adefovir dipivoxil; peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Adefovir dipivoxil
Drug: Peginterferon-alfa-2A
Drug: Ribavirin
Procedure: Liver Biopsy

SUMMARY:
This study will investigate the safety and effectiveness of using adefovir dipivoxil (ADV), pegylated interferon (PEG-INF), and ribavirin (RBV) in patients triple-infected with hepatitis B virus (HBV), hepatitis C virus (HCV), and HIV. Patients in this study must be taking lamivudine (3TC).

DETAILED DESCRIPTION:
The emergence of liver disease in HIV infected patients with coinfections of HBV and/or HCV has become increasingly important in disease progression in the post-HAART (highly active antiretroviral therapy) era. The overall rate of HBV and HCV infection in HIV infected persons is 5% to 10%. There is convincing evidence that HIV infection exacerbates the severity of viral hepatitis and the progression of liver disease. Hepatitis treatment studies have generally excluded HIV patients with both HBV and HCV. As such, the influence of HBV on HCV treatment in HIV infected patients is unknown. This study will investigate the safety and anti-HBV efficacy of ADV + PEG-INF + RBV triple therapy in patients with HCV, HIV, and 3TC-resistant HBV. The study will also evaluate the effect of HBV and HBV therapy on HCV and HIV disease progression.

Patients with documented HIV, 3TC-resistant HBV, and HCV will be randomized to one of two treatment regimens for 48 weeks. Patients in both groups will receive daily oral RBV and weekly subcutaneous injections of PEG-INF. Patients in Group A will receive daily ADV; patients in Group B will receive placebo. After 48 weeks of study treatment, all study medications will be discontinued and patients will undergo liver biopsy. Patients will then be followed for an additional 24 weeks. Throughout the study, investigators will monitor numerous lab values and patients will be asked to complete multiple adherence questionnaires. Subjects who have a confirmed 2 point increase in Child-Pugh-Turcotte liver disease prognosis score at any time during the study will permanently discontinue PEG-INF and RBV and register to Step 2 to receive open label ADV.

ELIGIBILITY:
Inclusion Criteria

* HIV positive
* Documented HCV viremia within 48 weeks prior to study entry
* HBV DNA >= 500,000 copies/ml within 12 weeks prior to study entry
* Chronic viral liver disease as documented by liver biopsy within 52 weeks prior to study entry
* Treated with 3TC for at least 26 weeks prior to study entry
* CD4+ count >200 cells/mm3 within 35 days prior to study entry
* HIV-1 viral load of <55,000 copies/ml within 35 days prior to entry
* Either have been on stable antiretroviral therapy for at least 12 weeks prior to study entry and plan to remain on same antiretroviral therapy OR have not received any antiretroviral therapy in the 12 weeks prior to the study and do not plan to begin antiretroviral therapy during the first 12 weeks of the study
* Acceptable methods of contraception

Exclusion Criteria

* History of any medical condition associated with chronic liver disease other than viral hepatitis
* History of ALT elevations over 3 X baseline level
* Child-Pugh-Turcotte (CPT) score > 5
* Previous suicide attempt or hospitalization for psychiatric illness within 2 years prior to study entry
* History of hypersensitivity to RBV, interferon, or other components of study medications
* Uncontrolled seizure disorder
* Certain medical conditions, including hepatitis D, autoimmune disorders, Chronic Obstructive Pulmonary Disease, cardiac disease, cancer, hemoglobinopathy, major organ transplant, kidney disease, opportunistic infection, and retinopathy
* Certain medications
* Pregnancy or breast-feeding
* Male partners of women who are pregnant
* Active drug or alcohol use or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dickens Theodore, M.D., Ph.D., Study Chair — University of North Carolina, Chapel Hill; Kenneth E Sherman, M.D., Ph.D, Study Chair — University of Cincinnati

REFERENCES:
- [Background] Benhamou Y, Bochet M, Thibault V, Calvez V, Fievet MH, Vig P, Gibbs CS, Brosgart C, Fry J, Namini H, Katlama C, Poynard T. Safety and efficacy of adefovir dipivoxil in patients co-infected with HIV-1 and lamivudine-resistant hepatitis B virus: an open-label pilot study. Lancet. 2001 Sep 1;358(9283):718-23. doi: 10.1016/s0140-6736(01)05840-8. PMID 11551579
- [Background] Soriano V, Garcia-Samaniego J, Bravo R, Gonzalez J, Castro A, Castilla J, Martinez-Odriozola P, Colmenero M, Carballo E, Suarez D, Rodriguez-Pinero FJ, Moreno A, del Romero J, Pedreira J, Gonzalez-Lahoz J. Interferon alpha for the treatment of chronic hepatitis C in patients infected with human immunodeficiency virus. Hepatitis-HIV Spanish Study Group. Clin Infect Dis. 1996 Sep;23(3):585-91. doi: 10.1093/clinids/23.3.585. PMID 8879784
- [Background] Xiong X, Flores C, Yang H, Toole JJ, Gibbs CS. Mutations in hepatitis B DNA polymerase associated with resistance to lamivudine do not confer resistance to adefovir in vitro. Hepatology. 1998 Dec;28(6):1669-73. doi: 10.1002/hep.510280629. PMID 9828233
- [Background] McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, Goodman ZD, Ling MH, Cort S, Albrecht JK. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med. 1998 Nov 19;339(21):1485-92. doi: 10.1056/NEJM199811193392101. PMID 9819446